CLINICAL TRIAL: NCT05387109
Title: An Exploratory Study of Penpulimab Combined With Anlotinib in Neoadjuvant Treatment of Resectable Stage II-IIIB Non-small Cell Lung Cancer
Brief Title: Penpulimab Combined With Anlotinib in Neoadjuvant Treatment of Resectable Non-small Cell Lung Cancer
Acronym: pcwaintrl
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQXB-L-II-001
Record Dates: First submitted 2022-04-18; First posted 2022-05-24 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: NSCLC
MeSH Terms: interventions — anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- penpulimab combined with anlotinib (Experimental): penpulimab: fixed dose of 200 mg, administered on the first day of each cycle, repeated every 3 weeks; Anlotinib: 12 mg, administered on days 1-14, orally once a day, about half an hour before breakfast (the daily dose should be as much as possible), taken with warm water, and repeated every 3 weeks
  Interventions: Drug: penpulimab combined with anlotinib

INTERVENTIONS:
Drug: penpulimab combined with anlotinib — penpulimab: fixed dose of 200 mg, administered on the first day of each cycle, repeated every 3 weeks; Anlotinib: 12 mg, administered on days 1-14, orally once a day, about half an hour before breakfast (the daily dose should be as much as possible), taken with warm water, and repeated every 3 weeks

SUMMARY:
Neoadjuvant therapy with penpulimab combined with anlotinib;with surgery within 4-6 weeks after drug withdrawal;Adjuvant therapy within 4-12 weeks after surgery

DETAILED DESCRIPTION:
1. Neoadjuvant therapy with penpulimab combined with anlotinib penpulimab: fixed dose of 200 mg, administered on the first day of each cycle, repeated every 3 weeks; Anlotinib: 12 mg, administered on days 1-14, orally once a day, about half an hour before breakfast (the daily dose should be as much as possible), taken with warm water, and repeated every 3 weeks.
2. operation treatment: Each subject will receive 3 cycles of study treatment, with surgery within 4-6 weeks after drug withdrawal.
3. Suggested dosing regimen in the adjuvant therapy phase:

It is recommended to give patients corresponding adjuvant therapy after surgery, and the specific adjuvant therapy plan will be formulated by the investigator according to the individual situation of the patient. The postoperative adjuvant therapy in this protocol is for reference only: complete pre-dose examination within 4-12 weeks after surgery, and conduct pre-administration evaluation of adjuvant therapy; use platinum-based chemotherapy (cisplatin: 75mg/m2, d1, Q3W, 4 cycles; in combination with docetaxel: 75mg/m2, d1, Q3W, 4 cycles, or in combination with pemetrexed: 500mg/m2, d1, Q3W, 4 cycles (for non-squamous cell carcinoma only) row 4 cycle of adjuvant therapy; then continued adjuvant single-agent penicillimab (200 mg, day 1, Q3W) for 1 year or until disease progression.

If the following conditions occur during the treatment, such as the subject's disease progression, drug toxicity and side effects intolerable, withdrawal of informed consent, etc., the patient will terminate the treatment. During the trial, the efficacy indicators and safety indicators were observed.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 years old ≤ age ≤ 70 years old, male or female;
* 2. ECOG score 0~1 points;
* 3. Patients with non-small cell lung cancer diagnosed by pathology (histology or cytology) (according to WHO 2015 classification);
* 4. Patients with positive PD-L1 expression (PD-L1≥1%);
* 5. According to the eighth edition of clinical tumor TNM staging, the subjects are patients with resectable stage II-IIIB (IIIB only T3N2) non-small cell lung cancer;
* 6. Have measurable lesions (according to RECIST 1.1 standard, the long diameter of CT scan of tumor lesions is ≥10mm, and the short diameter of CT scan of lymph node lesions is ≥15mm;);
* 7. Those who were initially diagnosed with non-small cell lung cancer before enrollment and had not undergone radiotherapy, chemotherapy, surgery and targeted therapy;
* 8. The subject must have sufficient cardiopulmonary function for the intended lung resection;
* 9. The function of major organs is normal, that is, the following criteria are met:

  1. Routine blood examination must meet the following requirements (no blood transfusion, no hematopoietic factor and no drug correction within 14 days):

     1. ANC ≥1.5×109/L;
     2. PLT ≥ 100×109/L;
     3. HB ≥ 90 g/L;
  2. The biochemical examination must meet the following standards:

     1. TBIL≤1.5×ULN;
     2. ALT, AST≤2.5×ULN
     3. Serum creatinine sCr≤1.5×ULN, endogenous creatinine clearance rate≥50mL/min (Cockcroft-Gault formula);
     4. ALB ≥30 g/L
  3. Coagulation function must meet: INR≤1.5×ULN and APTT≤1.5×ULN;
* 10. Normal lung function or mild to moderate abnormality, and can tolerate surgery;

  1. VC%>60%
  2. FEV1>1.2L, FEV1%>40%
  3. DLco>40%
* 11. Female subjects of childbearing age must undergo a serum pregnancy test within 3 days before starting the study drug, and the result is negative, and are willing to use a medically approved high-efficiency contraceptive during the study and within 3 months after the last dose of the study drug Measures (eg: IUD, contraceptives, or condoms); for male subjects whose partners are females of childbearing age, surgical sterilization, or consent to use an effective method of contraception.

Exclusion Criteria:

* 1. Target disease exclusion criteria

  1) Subjects who have previously received anti-PD-1 (L1) or CTLA4 monoclonal antibody therapy;
* 2. Medical history and comorbidities

  1. Suffering from other malignant tumors in the past 3 years;
  2. Suffering from any active autoimmune disease or history of autoimmune disease (as follows, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, Hypothyroidism (may be included after hormone replacement therapy); patients with vitiligo or childhood asthma in complete remission and without any intervention as adults may be included; patients requiring medical intervention with bronchodilators are not included;
  3. The use of immunosuppressive drugs within 14 days before the first use of the study drug, excluding nasal spray and inhaled corticosteroids or systemic steroids at physiological doses (ie, no more than 10 mg/day prednisone or its equivalent) );
  4. Uncontrolled hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg despite optimal medical treatment);
  5. Newly diagnosed angina pectoris within 3 months before screening or myocardial infarction within 6 months before screening; arrhythmia (including QTcF: ≥450 ms in males, ≥470 ms in females) requires long-term use of antiarrhythmic drugs and New York Cardiac Association classification ≥ class II cardiac insufficiency; or uncontrolled heart failure;
  6. There is evidence of past or current pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiological pneumonia, drug-induced pneumonia, and severely impaired lung function;
  7. Complicated severe infection within 4 weeks before the first dose (eg: need for intravenous infusion of antibiotics, antifungal or antiviral drugs), or unexplained fever >38.5°C during the screening period/before the first dose;
  8. Clinically significant hemoptysis (more than 50 mL of hemoptysis per day) within 3 months before the study, or clinically significant bleeding symptoms or obvious bleeding tendency (such as gastrointestinal bleeding, gastric ulcer bleeding, gastrointestinal bleeding, hemorrhagic gastric Ulcer, fecal occult blood++ or above baseline, or suffering from vasculitis, etc.).
  9. Active bleeding or abnormal coagulation function (INR>2.0, PT>16s), with bleeding tendency or receiving thrombolysis, anticoagulation or antiplatelet therapy;
  10. Renal insufficiency: urine routine indicates urine protein ≥ ++, or confirmed 24-hour urine protein amount ≥ 1.0g;
  11. Imaging shows that the tumor has invaded around important blood vessels or the investigator judges that the patient's tumor has a high possibility of invading important blood vessels during treatment and causing fatal hemorrhage;
  12. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
  13. Administer live attenuated vaccines within 4 weeks before the first dose or plan during the study period;
  14. Patients with central squamous cell carcinoma diagnosed by imaging examination and pathological examination;
* 3. Physical examination and laboratory findings

  1. Patients with congenital or acquired immunodeficiency, such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (positive hepatitis C antibody, and high HCV-RNA) (the lower limit of detection of the analytical method) or co-infection with hepatitis B and C;
  2. Pregnant or breastfeeding women; patients with childbearing potential who are unwilling or unable to take effective contraceptive measures;
  3. Those who are known to be positive for EGFR/ALK gene mutation, and those whose EGFR/ALK gene mutation status is unknown are not required to be tested;
* 4. Allergies, anaphylaxis and adverse drug reactions

  1. Severe allergic reactions to other monoclonal antibodies;
  2. Allergy or intolerance to infusion;
  3. Have a history of severe allergy to Anlotinib or its preventive medicines;
* 5. Subjects who are participating in other clinical studies or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or 5 half-lives of the research drug;
* 6. The subject is known to have a history of psychotropic substance abuse, alcohol or drug abuse; The investigator believes that there are any conditions that may harm the subject or prevent the subject from meeting or performing the research requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-04-20 (Estimated); Study Completion 2024-04-20 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response, pCR | 12months
  To evaluate the pathological complete response rate (pCR) of pembrolizumab combined with anlotinib neoadjuvant therapy for resectable non-small cell lung cancer.

SECONDARY OUTCOMES:
Major pathologic response, MPR | 12months
  Evaluate the major pathologic response rate (MPR)
Disease free survival,DFS | 12months
  defined as, according to the RECIST1.1 criteria, the time between subjects from enrollment to disease recurrence or death (for any reason)

CONTACTS AND LOCATIONS:
Overall Officials: Tao Jiang, Study Chair — Tang-Du Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] NCCN Clinical Practice Guidelines in Oncology (NCCN Guidelines®) Non-small Cell Lung Cancer Version 2.2016.
- [Result] McElnay P, Lim E. Adjuvant or neoadjuvant chemotherapy for NSCLC. J Thorac Dis. 2014 May;6 Suppl 2(Suppl 2):S224-7. doi: 10.3978/j.issn.2072-1439.2014.04.26. PMID 24868440
- [Result] Forde PM, Chaft JE, Smith KN, Anagnostou V, Cottrell TR, Hellmann MD, Zahurak M, Yang SC, Jones DR, Broderick S, Battafarano RJ, Velez MJ, Rekhtman N, Olah Z, Naidoo J, Marrone KA, Verde F, Guo H, Zhang J, Caushi JX, Chan HY, Sidhom JW, Scharpf RB, White J, Gabrielson E, Wang H, Rosner GL, Rusch V, Wolchok JD, Merghoub T, Taube JM, Velculescu VE, Topalian SL, Brahmer JR, Pardoll DM. Neoadjuvant PD-1 Blockade in Resectable Lung Cancer. N Engl J Med. 2018 May 24;378(21):1976-1986. doi: 10.1056/NEJMoa1716078. Epub 2018 Apr 16. PMID 29658848
- [Result] Rusch V W, Chaft J E, Johnson B, et al. Neoadjuvant atezolizumab in resectable non-small cell lung cancer (NSCLC): Initial results from a multicenter study (LCMC3)[J]. Journal of Clinical Oncology, 2018, 36, 8541. DOI: 10.1200/JCO. 2018.36.15_suppl.8541.
- [Result] Cascone T, William W N, Weissferdt A, et al. LBA49 Neoadjuvant nivolumab (N) or nivolumab plus ipilimumab (NI) for resectable non-small cell lung cancer (NSCLC)[J]. Annals of Oncology, 2018, 29(suppl_8): mdy424. 059.
- [Result] Provencio-Pulla M, Nadal-Alforja E, Cobo M, et al. Neoadjuvant chemo/immunotherapy for the treatment of stages IIIA resectable non-small cell lung cancer (NSCLC): A phase II multicenter exploratory study-NADIM study-SLCG [J]. Journal of Clinical Oncology, 2018, 36, 8521. DOI: 10.1200/JCO. 2018.36.15_suppl.8521.
- [Result] Jonathan Spicer, Changli Wang, Fumihiro Tanaka, et al. Surgical outcomes from the phase 3 CheckMate 816 trial: Nivolumab (NIVO) + platinum-doublet chemotherapy (chemo) vs chemo alone as neoadjuvant treatment for patients with resectable non-small cell lung cancer (NSCLC) [J]. 2021, ASCO, abstract 8503.
- [Result] Zhao X, Su Y, You J, Gong L, Zhang Z, Wang M, Zhao Z, Zhang Z, Li X, Wang C. Combining antiangiogenic therapy with neoadjuvant chemotherapy increases treatment efficacy in stage IIIA (N2) non-small cell lung cancer without increasing adverse effects. Oncotarget. 2016 Sep 20;7(38):62619-62626. doi: 10.18632/oncotarget.11547. PMID 27566586
- [Result] Chaft JE, Rusch V, Ginsberg MS, Paik PK, Finley DJ, Kris MG, Price KA, Azzoli CG, Fury MG, Riely GJ, Krug LM, Downey RJ, Bains MS, Sima CS, Rizk N, Travis WD, Rizvi NA. Phase II trial of neoadjuvant bevacizumab plus chemotherapy and adjuvant bevacizumab in patients with resectable nonsquamous non-small-cell lung cancers. J Thorac Oncol. 2013 Aug;8(8):1084-90. doi: 10.1097/JTO.0b013e31829923ec. PMID 23857398
- [Result] Mislang A, Coward J, Cooper A, et al. 157P Efficacy and safety of penpulimab (AK105), a new generation anti-programmed cell death-1 (PD-1) antibody, in upper gastrointestinal cancers [J]. Annals of Oncology, 2020, 31.
- [Result] Kotasek D, Coward J, Souza P, et al. A phase I dose escalation and dose expansion study of the anti-programmed cell death-1 (PD-1) antibody AK105 [J]. Journal of Clinical Oncology, 2019, 37(15_suppl): e14006-e14006.
- [Result] Song Y, Zhu J, Lin N, et al. A phase I/II study of the anti-programmed cell death-1 (PD-1) antibody AK105 in patients with relapsed or refractory classic Hodgkin lymphoma (cHL) [J]. Journal of Clinical Oncology, 2019, 37(15_suppl): e19017-e19017.